CLINICAL TRIAL: NCT03836950
Title: rTMS as a Cognitive Rehabilitation Approach in Veterans With Parkinson'sDisease
Brief Title: rTMS to Improve Cognition in Parkinson's
Acronym: TMSCogReP
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: VA Office of Research and Development (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: N2938-W; IK2RX002938 (NIH); 2023CWR-NDS-831171250 (Other Grant/Funding Number: Cures Within Reach)
Record Dates: First submitted 2019-01-28; First posted 2019-02-11 (Actual); Last update posted 2025-09-05 (Actual); Status verified 2025-09

CONDITIONS: Parkinson's Disease; Mild Cognitive Impairment
Keywords: rTMS; Parkinson's disease; mild cognitive impairment; executive function; neuromodulation; functional connectivity
MeSH Terms: conditions — Parkinson Disease; Cognitive Dysfunction

STUDY DESIGN:
Intervention Model Description: randomized control trial. Participants will receive either active or sham rTMS
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- active rTMS (Experimental): For active rTMS, a butterfly coil and MagVenture MagProX100 stimulator (MagVenture, Falun, Denmark) will be used. One rTMS session will consist of 40 trains of 5sec each at 110% of resting motor threshold and 15Hz will be provided at the left DLPFC.
  Interventions: Device: MagVenture MagProX100 stimulator (MagVenture, Falun, Denmark)
- sham rTMS (Sham Comparator): For sham rTMS, the procedure will be carried out at the left DLPFC but a sham coil will be used. The MagVenture coil has an active side and a placebo side allowing a double-blind study to be conducted. The sham system looks, sounds and feels like active rTMS.
  Interventions: Device: MagVenture MagProX100 stimulator (MagVenture, Falun, Denmark)

INTERVENTIONS:
Device: MagVenture MagProX100 stimulator (MagVenture, Falun, Denmark) — The coil will be held tangentially to the skull at approximately 45º from the midline. One rTMS session will consist of 40 trains of 5sec each at 110% of resting motor threshold and 15Hz will be provided at the left DLPFC.
  Arms: active rTMS
Device: MagVenture MagProX100 stimulator (MagVenture, Falun, Denmark) — The coil will be held tangentially to the skull at approximately 45º from the midline. The sham coil will not release any stimulation, but it will look, feel and sound like the real rTMS
  Arms: sham rTMS

SUMMARY:
The purpose of this study is to examine safety, feasibility, and the behavioral and brain effects of a non-invasive treatment, repetitive transcranial magnetic stimulation (rTMS), for Veterans with Parkinson's disease or atypical parkinsonism and mild impairments in their thinking. The hypothesis is that rTMS can improve thinking for people with Parkinson's disease or atypical parkinsonism who are experiencing mild problems with their thinking ability.

DETAILED DESCRIPTION:
Repetitive transcranial magnetic stimulation (rTMS) shows promise as an effective cognitive neurorehabilitation treatment. To date, no rTMS studies have assessed the effect of rTMS on cognitive function in PD-MCI. Nor has there been PD neurophysiological studies using rTMS to examine neural plasticity in cognitive neural networks. This study seeks to fill this gap by conducting a small scaled pilot randomized controlled trial (RCT) designed to assess the safety and therapeutic effects of rTMS on cognitive outcomes as well as on brain connectivity in Veterans with PD-MCI. PD-MCI participants will be randomized to either active rTMS or sham rTMS. Participants will complete a standardized neurocognitive battery assessment at baseline, endpoint and at a one month follow-up. The primary outcome is change in executive function. Secondary outcomes include performance on other cognitive domain tasks and a proximal measure of real-life function that captures relevant functional changes related to cognitive impairment in PD. Multi-modal neuroimaging, in a subsample of participants, will be used to study neural connectivity changes induced by rTMS. Changes in resting state functional connectivity, grey matter volume via voxel-based morphometry and white matter integrity via diffusion tensor imaging will be assessed at baseline and endpoint. To inform how to optimize rTMS treatment in PD-MCI, these changes will be correlated with changes in cognitive performance.

ELIGIBILITY:
Inclusion Criteria:

* Veterans who seek services at Hines VA Hospital or Jesse Brown VA Medical Center
* Diagnosis of PD or atypical parkinsonism as determined by a neurologist
* Meet criteria for having mild cognitive impairment
* Receiving stable (i.e., no changes in medication and medication dose) medication and who are expected to remain on stable medication for the duration of the RCT
* Speak and read English
* 50 years or older

Exclusion Criteria:

* Dementia
* Failure to demonstrate decision making capacity
* History of deep brain stimulation surgery
* Severe depression
* Resting head tremor
* Dyskinesia that will interfere with collecting imaging data
* Has congestive heart failure
* Implanted cardiac pacemaker or defibrillator
* Cochlear implant, nerve stimulator, or intracranial metal clips
* Implanted medical pump
* Increased intracranial pressure
* History of claustrophobia
* Metal in eyes/face, shrapnel/bullet remnants in brain
* Participants at potential increased risk of seizure including those who have the following:

  * history (or family history) of seizure or epilepsy
  * history of stroke, head injury, or unexplained seizures
  * presence of other neurological disease that may be associated with an altered seizure threshold

    * such as CVA, cerebral aneurysm, dementia, increased intracranial pressure
* Concurrent medication use such as tricyclic antidepressants, neuroleptic medications, any other drug known to lower seizure threshold
* Secondary conditions that may significantly alter electrolyte balance or lower seizure threshold
* No quantifiable motor threshold such that rTMS dosage cannot be accurately deter-mined

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 56 (Estimated)
Dates: Start 2020-04-01 (Actual); Primary Completion 2026-03-31 (Estimated); Study Completion 2027-03-30 (Estimated)

PRIMARY OUTCOMES:
change in NIH sponsored Executive Abilities: Measures and Instruments for neurobehavioral evaluation and re-search (NIH-EXAMINER) executive composite score | baseline, 8 weeks, 12 weeks
  The NIH-EXAMINER has an established 3-factor model defined by (1) cognitive control, (2) working memory (3) fluency. A confirmatory factor analysis indicates these 3-factors load on to 1-factor: executive composite score. Seven tests in the NIH-EXAMINER will be used to compute the composite score

CONTACTS AND LOCATIONS:
Overall Officials: Sandra L. Kletzel, PhD BA, Principal Investigator — Edward Hines Jr. VA Hospital, Hines, IL
Locations (2):
- United States (2):
  - Jesse Brown VA Medical Center, Chicago, IL, Chicago, Illinois
  - Edward Hines Jr. VA Hospital, Hines, IL, Hines, Illinois

IPD SHARING:
Plan to Share IPD: Yes
Raw and/or normalized data will be made available in the form of Excel files. MRI images will anonymized and made available through the Northwestern University Neuroimaging Data Archive (NUNDA).
Time Frame: Final data sets will be made available as per Hines VA Hospital local policy for long term storage and access until enterprise-level resources become available.
Access Criteria: These data will be available upon request by researchers and scientists in accordance with federal guidelines and Hines local policy.